CLINICAL TRIAL: NCT07306962
Title: Does Computer-assist Virtual Lesion Segmentation Ushers to a Change in the Literature Consensus Regarding Mandibular Ameloblastoma Radiographic Safety Margin?. A Clinical Case Series
Brief Title: Virtual Lesion Segmentation and Mandibular Ameloblastoma Radiographic Safety Margin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-12-25/SM-Amelo
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Ameloblastoma
Keywords: segmental mandibular defect; anterior iliac crest; virtual surgical planning accuracy
MeSH Terms: conditions — Ameloblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual lesion segmentation for mandibular ameloblastoma (Experimental): Patient with mandibular ameloblastoma managed with virtual surgical planning & Virtual lesion segmentation for the determination of a radiographic 10-mm safety margin.
  Interventions: Device: Virtual lesion segmentation for mandibular ameloblastoma

INTERVENTIONS:
Device: Virtual lesion segmentation for mandibular ameloblastoma — Patient with mandibular ameloblastoma managed with virtual surgical planning & Virtual lesion segmentation for the determination of a radiographic 10-mm safety margin.

SUMMARY:
Reconstruction of segmental mandibular defects is in a continuous state of evolution utilizing the recent advances in Computer-Aided Designing (CAD) and preoperative Virtual Surgical Planning (VSP). The anterior iliac crest is one of the ideal reservoirs for autogenous harvesting of a bi-cortical bone block with 1:1 cortical to cancellous bone ratio which is optimal for rapid and predictable consolidation. The aim of this study is the utility of VSP guided by CT and confirmation by histopathological analysis in achieving negative margins and preventing recurrence of mandibular ameloblastoma.

DETAILED DESCRIPTION:
A total of 10 patients having segmental mandibular defects will be selected. All defects will be reconstructed using anterior iliac crest in utilizing preoperative virtual surgical planning and intraoperative resection and reconstruction guides. The resected mandible will be evaluated by radiographic three-dimensional that will be performed to determine the accuracy of the VSP guided by CT, along with histopathological analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed ameloblastoma using a preoperative biopsy.
2. Patients with ameloblastoma that require segmental mandibular continuity defect, not involving the condyle.

Exclusion Criteria

1. Patients with lateral segmental mandibular defect involving the condyle.
2. Patients with an active infection at the site of resection.
3. Patients with recurrent lesion after resection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Histological analysis and degree of lesion invasion determination | 1 month
  The specimen with the the mounted Safety Margin Calibration Guide will be sent for histological evaluation. For light microscopic examination, the specimens will be embedded in paraffin wax blocks after being fixed in 10% formalin, neutrally buffered, cleaned, and dehydrated using increasing ethanol concentrations. Tissue sections will be cut to a thickness of 4 μm, and stained with hematoxylin and eosin to be examined under a light microscope.
  The specimen will be cut, using the S35 (0.254-mm thickness) microtome blade, at the preoperatively determined margins according to the virtual lesion segmentation from the proximal and distal sides of the lesion. Since the study is limited to segmental mandibular resection, the full lower border of the mandible was resected and their will be no need for assessment of either coronal or apical margins

SECONDARY OUTCOMES:
Postoperative resection margin accuracy analysis | 1 week
  At the end of the surgical procedure, the Safety margin caliberation guide was mounted on the specimen and fixed using 2 2.0-mm miniscrews. A radiographic MSCT scan for the resected mandible with the Safety margin caliberation guide will be obtained using same preoperative scanning parameters. The DICOM data of the scanned Specimen will be segemented to create an Actual Resected Specimen Model (ARSM). The RSM will be superimposed with the preoperative Virtual Resected Specimen Model (VRSM) using the miniscrews as radiographic markers for superimposition. The postoperative accuracy of the virtually assisted surgery will be conducted using the 3D-analysis software (GOM-Inspect software*) For each of the selected 2D and 3D parameters, the Deviation will be calculated by subtracting the ARSM values from the VRSM. The absolute mean (Δ) for all of the operated patients will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: yehia A El-Mahallawy, PhD, Principal Investigator — Faculty of Dentistry, Alexandria University, Alexandria, Alexandria
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified to protect the participant data. patients signed an informed consent for the use of their medical records and data for study.